CLINICAL TRIAL: NCT01253499
Title: A Phase 1 Study Consisting of a Double-Blind, Placebo Controlled Multiple Dose Study of TRx0037 in Healthy Elderly Volunteers
Brief Title: Multiple Dose Study of TRx0037
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TauRx Therapeutics Ltd (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Professor Claude M. Wischik, Chairman, TauRx Therapeutics Ltd
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: TRx-037-003
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (1):
- TRx0037 (Experimental): Double blind placebo controlled study of TRx0037 in healthy elderly volunteers to assess safety, tolerability, bioavailability and pharmacokinetics
  Interventions: Drug: TRx0037

INTERVENTIONS:
Drug: TRx0037 — 75mg and 100mg tablets used to create doses of 100mg and 175mg. Active placebo 2mg and blank placebo used as comparators.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of TRx0037 after multiple doses in elderly volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female 55 and over
* No clinically important abnormal physical finding
* No clinically significant lab results
* Normal ECG
* Normal BP and HR
* BMI between 19 and 32
* Weight 50 to 100 kg
* Able to communicate
* Provide written informed consent
* Non smokers
* Males to use contraception
* Females to be surgically sterile or post menopausal

Exclusion Criteria:

* Administration of any IMP other than study drug within 12 weeks before entry
* Use of any prescribed meds, St John's wort, over the counter meds as described in the protocol
* Surgical or medical condition that might interfere with IMP
* History of drug or alcohol abuse
* Clinically significant allergy requiring treatment
* Loss of greater than 400ml of blood within 12 weeks.
* Serious adverse reaction or hypersensitivity to any drug
* Presence of Hep B, Hep c or HIV-1 or HIV-2 at screening
* Presence of G6PD at screening
* History of methaemoglobinaemia
* Partner who is pregnant of lactating
* Positive Pregnancy test

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Bioavailability | 19 Days (7-10 day follow up)
  The bioavailability of TRx0037 in an older population closer to the typical age range of the target patient population.
Pharmacokinetics | 19 Days (7-10 day follow up)
  The pharmacokinetics for single doses of TRx0037 in healthy elderly volunteers.
Safety and tolerability | 19 Days (7-10 day follow up)
  Safety and tolerability measurements including adverse events, physical examination findings, vital signs, ECG, and clinical laboratory measurements for single doses of TRx0037

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Dr Mair, MBChB, Principal Investigator — Quotient Clinical